CLINICAL TRIAL: NCT02060656
Title: A Randomised Phase II Study Comparing LEnalidomide Plus Rituximab, GEmcitabine and Methylprednisolone (LR-GEM) to Rituximab, Gemcitabine, Methylprednisolone and cisplatiN (R-GEM-P) in Second-line Treatment of Diffuse Large B-cell Lymphoma (DLBCL).
Brief Title: Phase II Study Comparing LR-GEM to R-GEM-P in Second-line Treatment of Diffuse Large B-cell Lymphoma (LEGEND)
Acronym: LEGEND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMH CCR: 3862; 2012-002620-32 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-02-12 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Relapsed or refractory Diffuse Large B-Cell Lymphoma after R-CHOP chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Gemcitabine; Methylprednisolone; Rituximab; Cisplatin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control: R-GEM-P (Active Comparator): Rituximab,Gemcitabine, Methylprednisolone,Cisplatin.
  Interventions: Drug: Gemcitabine; Drug: Methylprednisolone; Drug: Rituximab; Drug: Cisplatin
- Experimental: LR-GEM (Experimental): Lenalidomide, Rituximab, Gemcitabine, Methylprednisolone
  Interventions: Drug: Gemcitabine; Drug: Methylprednisolone; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 IV D1, D8, D15 every 28 days
Drug: Methylprednisolone — 1000mg/m2 IV or PO D1-5 every 28 days
Drug: Rituximab — 375mg/m2 IV D1, D15 every 28 days
Drug: Cisplatin — 100mg/m2 IV D15 every 28 days
  Arms: Control: R-GEM-P
Drug: Lenalidomide — 25mg PO D1-21 every 28 days
  Arms: Experimental: LR-GEM

SUMMARY:
This is a randomised, phase II open-labelled two-arm study comparing R-GEM-P and LR-GEM in second-line treatment of Diffuse Large B-cell lymphoma. Eligible patients will be randomised 1:1 between R-GEM-P and LR-GEM.

DETAILED DESCRIPTION:
Objectives:

Primary

To assess the complete response rate to LR-GEM (lenalidomide, rituximab, gemcitabine and methylprednisolone) and R-GEM-P (rituximab, gemcitabine,cisplatin and methylprednisolone) following 3 cycles of induction treatment as secondline therapy for patients with Diffuse Large B-cell Lymphoma.

To investigate in both arms:

* Overall response rate following 3 cycles of induction treatment evaluated by IWG 2007 criteria
* Event-free survival
* Overall survival
* Rate of successful stem cell harvest
* Toxicity
* Subgroup analyses will be performed on the primary endpoint by cell-of-origin immunohistochemical subtype using the Choi method[2] (GCB vs non-GCB), morphological subtype (centroblastic vs immunoblastic vs other), IPI (0-1 vs ³2),and previous response to treatment (£12 vs > 12 months), and eligibility for ASCT at randomisation.

Treatment:

LR-GEM: lenalidomide plus rituximab, gemcitabine and methylprednisolone every 28 days. R-GEM-P: rituximab, gemcitabine, methylprednisolone and cisplatin every 28 days.

Assessment Schedule:

* Patients will be reviewed at baseline and prior to each scheduled dose of treatment for toxicity
* Radiological tumour assessment will be done with contrast-enhanced CT scan after the 1st and 3rd cycles in both arms.
* PET/CT scan will be performed at baseline and upon completion of induction treatment (3-4 weeks after last dose of chemotherapy). If PET/CT scan is performed with a contrast-enhanced CT, then patients do not need a separate CT scan.
* Follow up after completion of induction treatment will be at 3 monthly intervals for the first 12 months in Arm A and at monthly intervals for the first 12 months for patients in Arm B. Thereafter follow up in both Arm A and B will be at 6 monthly intervals for 2 years, then annually up until 5 years in total.
* CT scan at 3 & 12 months post induction treatment in both arms
* Following disease progression patients will be followed for survival every 3 months until death

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD20+ Diffuse Large B-Cell Lymphoma
* Availability of a tumour block containing adequate histological material for central pathology review, establishment of morphological and ontogenic subtype.
* Surgically acquired tissue samples are preferred but if core biopsy is the only suitable means by which to acquire a tissue sample then it is suggested than at least 2 cores are taken so that one can be embedded and sent for central review and one retained locally.
* Relapsed after or refractory to one prior line of chemotherapy for DLBCL containing both rituximab and an anthracycline. Relapsed is defined as investigator assessed progression after first line treatment. Refractory is defined as patients who progressed during or who did not achieve complete remission with first line treatment (which should include radiotherapy if the patient had localised refractory disease)
* Eligible for combination chemotherapy regimen.
* Patient is 18 years of age on the day of signing informed consent.
* ECOG performance status 0, 1 or 2.
* Baseline PET or CT scans must demonstrate FDG avid disease compatible with CT defined anatomical tumour sites.
* Adequate bone marrow function: absolute neutrophil count (ANC) 1.0x109/l, white blood cell count 3x109/l, platelets 100x109/l, haemoglobin (Hb) 9g/dl (can be post-transfusion), unless deemed disease related
* Adequate renal function: calculated creatinine clearance 40ml/minute.
* Adequate liver function: serum bilirubin 1.5x ULN, ALT/AST 2.5x ULN, ALP 3x ULN (in the absence of liver metastases). If liver metastases are present, ALT, AST or ALP 5x ULN are permitted. Isolated hyperbilirubinaemia due to Gilbert's disease is acceptable.
* Female patient of childbearing potential (FCBP) must have two negative serum β-hCG pregnancy tests at baseline.
* FCBP agreeable to practice complete and true sexual abstinence or use two forms of contraception from 28 days prior to the period of study treatment and for 12 months after the last dose of study drugs.
* Male patients agreeable to practice complete and true sexual abstinence or use condoms from 28 days prior to the period of study treatment and for 12 months after the last dose of study drugs.
* Recovery from toxicity from previous anti-cancer treatment to grade 1.

Exclusion Criteria:

* Documented or symptomatic central nervous system involvement or leptomeningeal disease.
* Any other clinically significant disease or co-morbidity which may adversely affect the safe delivery of treatment within this trial, including active or chronic infection,poorly controlled diabetes mellitus, congestive cardiac failure, cardiac arrhythmia, coronary artery disease, cerebrovascular disease, or severe pulmonary disease.
* Any other malignancies diagnosed or treated within the last 5 years (other than curatively treated basal cell or squamous cell carcinoma of the skin and/or in situ carcinoma of the cervix or breast).
* Received drug treatment for cancer within 21 days of commencing study treatment.
* Received previous lenalidomide
* Evidence of human immunodeficiency virus infection, hepatitis C virus, acute or active hepatitis B infection.
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within one year of finishing study treatment.
* Hypersensitivity or contraindication to any of the study drugs as stated in the SmPCs for each of the study drugs.
* Prior stem cell or solid organ transplant
* Treatment with an investigational product within 30 days prior to enrollment
* Not able to provide fully informed consent because of intellectual impairment or psychiatric disorder
* Patient unwilling or not able to adhere to the Lenalidomide Pregnancy Prevention Programme.
* Treatment with combined oral contraceptive pill within 30 days prior to enrollment.
* Treatment with hormone replacement therapy within 30 days prior to enrollment
* Treatment with erythropoeitic agents within 30 days prior to enrollment
* Baseline hearing impairment, which in the opinion of the investigator, may significantly worsen with treatment with cisplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | Approximatley after 12 weeks of randomisation

SECONDARY OUTCOMES:
Overall Response Rate | Approximately 12 weeks after randamisation
Event-free Survival | This will be calculated from the date of randomisation until the date of treatment failure up to 104 weeks
Overall Survival | this will be calculated from the date of randomisation until the date of death, irrespective of its cause.
Rates of successful stem cell harvest | This will be calculated by the amount of stem cells collected and number of stem cell harvest attempts per patient up to 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust - London and Surrey, London, United Kingdom